CLINICAL TRIAL: NCT04233437
Title: Drug-Drug Interaction Study of MLC1501 Using Cocktail of Drugs Acting as Sensitive Clinical Probes/Substrates of Cytochrome P450 Isoenzymes and Transporters in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Moleac Pte Ltd. (Industry)
Collaborators: Moleac Australia Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SAFE2019_01
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to either CYP or Transporter cohort in ratio of 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CYP Cohort (Experimental): MLC1501 & CYP cocktail drugs
  Interventions: Drug: MLC1501; Drug: CYP Cocktail
- Transporter Cohort (Experimental): MLC1501 & Transporter cocktail drugs
  Interventions: Drug: MLC1501; Drug: Transporter Cocktail

INTERVENTIONS:
Drug: MLC1501 — MLC1501 capsules (4 capcules (2000 mg) twice a day)
Drug: CYP Cocktail — Repaglinide 0.25 mg, caffeine 100 mg, warfarin 10 mg (with vitamin K), omeprazole 40 mg, dextromethorphan 30 mg, midazolam 2 mg
  Arms: CYP Cohort
Drug: Transporter Cocktail — Digoxin 0.25 mg, furosemide 1 mg, metformin 10 mg, rosuvastatin 10 mg
  Arms: Transporter Cohort

SUMMARY:
This is a single-centre phase I study to assess the Drug-Drug Interaction potential of MLC1501 with a cocktail of drugs acting as sensitive clinical probe substrates of Cytochrome P450 isoenzymes and Transporters in healthy subjects .

The study will have 2 cohorts, one for the CYP study and the other for the Transporters study. Eligible subjects (n=24) will be assigned to one of the 2 cohorts in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, male or female
2. 18 to 55 years old
3. Body mass index of 18 to <30 kg/m2
4. Able to understand the study requirements and provide written informed consent for participation in the study.

Exclusion Criteria:

1. Any history of or presences of medical condition (such as hypertension, diabetes mellitus, hyperlipidaemia, or any cardiac, neurological, pulmonary, gastrointestinal, hepatic, hematologic, or renal disease).
2. Concurrent use of any medication to treat any medical condition

   * CYP cohort: Within 72hr of the first dose of repaglinide or 5 half-lives of dosing of any medication, whichever longer, and until the end of the study
   * Transporter cohort: Within 72hr of first dose of Transporter cocktail or 5 half-lives of dosing of any medication, whichever longer, and until the end of the study
3. Surgery within 4 weeks prior to Screening, as determined by the Investigator
4. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs including cholecystectomy (uncomplicated appendectomy and hernia repair will be allowed).
5. Use of tobacco- or nicotine-containing products within 72 hours prior to dosing.
6. Current substance or alcohol abuse/addiction
7. Women who are pregnant or breastfeeding.
8. Women who are of child-bearing potential unless they maintain abstinence during study period or use barrier method of contraception and male partner using condom. Systemically acting hormonal contraceptives are not allowed, however locally acting hormonal contraceptives i.e. intrauterine device (IUD) (including Mirena) is allowed. Menopausal/post-menopausal women without menstruation for 12 consecutive months or surgically sterilized women may also be included. Intake of oral contraceptive pills or hormone replacement therapy is not allowed.
9. Male subjects with female partner of child-bearing potential unless they maintain abstinence during study period or use of barrier method of contraception with female partner using any method of contraception.
10. Male subjects unless they are willing not to donate sperm 90 days from last study drug administration.
11. Use or intend to use any medications or products known to alter drug absorption, metabolism, or elimination processes, vitamin, minerals, herbal/traditional medicines including St John's Wort. 20 days prior to the first dose, unless deemed acceptable by the Investigator.
12. Caffeine-containing beverages, substance, alcohol, grapefruit juice/grapefruit containing products, Seville oranges/ juice/, chamomile, liquorice, broccoli or brussels sprouts within the 72hrs prior to dosing.
13. Any known hypersensitivity/allergic reaction/anaphylaxis to food, animal stings, drugs inclusive of drugs used in CYP and transporter cocktail in the study /components of MLC1501, or members of the Fabaceae/Leguminosae family (e.g. legume, pea, bean), Polygalaceae family (e.g. milkwort, snakeroot), Apiaceae/ Umbelliferae family (e.g. anise, caraway, carrot, celery, dill, parsley, parsnip), or Quillaja bark (soapbark).
14. Any abnormal physical examination findings or laboratory results (including serum electrolytes such as sodium, potassium and chloride) or abnormal ECG findings (like atrial fibrillation or flutter, supraventricular tachycardia, pre-excitation or wolff Parkinson white. Etc) at screening that is considered to be clinically significant by the study investigator.
15. Any medical condition which, in the study investigator's opinion, may jeopardize the subject by his/her participation in this study, may hamper his/her ability to complete procedures required in the study, or affect the validity of the study results.
16. Administration of an investigational drug (new chemical entity) or device trial within 90 days or 5 half-lives, whichever is longer, prior to the first dose, or concomitant participation in an investigation study involving no drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
Change in area under curve (AUC) of individual substrates is being assessed between cocktail alone and cocktail + MLC1501 administration | Through study completion, an average of 29 days and 18 days for CYP and Transporter cohort, respectively.
  Assayed in plasma samples collected at various time points after cocktail administration and cocktail + MLC1501 administration.
Change in maximum concentration (Cmax) of individual substrates is being assessed between cocktail alone and cocktail + MLC1501 administration | Through study completion, an average of 29 days and 18 days for CYP and Transporter cohort, respectively.
  Assayed in plasma samples collected at various time points after cocktail administration and cocktail + MLC1501 administration.
Change in time taken to reach maximum concentration (Tmax) of individual substrates is being assessed between cocktail alone and cocktail + MLC1501 administration | Through study completion, an average of 29 days and 18 days for CYP and Transporter cohort, respectively.
  Assayed in plasma samples collected at various time points after cocktail administration and cocktail + MLC1501 administration.

SECONDARY OUTCOMES:
Ratio of geometric means (GMR) between cocktail alone and cocktail + MLC1501 for the AUC and Cmax of the corresponding probe | Through study completion, an average of 29 days and 18 days for CYP and Transporter cohort, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia